CLINICAL TRIAL: NCT04500041
Title: Casting Vs Bracing for Idiopathic Early-Onset Scoliosis
Acronym: CVBT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Orthopedic Research and Education Foundation (Other); Pediatric Spine Study Group (Unknown)
Responsible Party: Principal Investigator, Stuart L. Weinstein, MD, Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202003169
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Scoliosis Idiopathic; Early-Onset Scoliosis Deformity of Spine
Keywords: Cast; Brace; Spinal Orthosis; Spinal Orthotic
MeSH Terms: interventions — Braces

STUDY DESIGN:
Intervention Model Description: Treatment (casting or bracing) via randomized assignment OR based on family preference
Who Masked: Outcomes Assessor
Masking Description: Study outcome is determined from serial radiographs. Radiographic readers will be blinded to the treatment assigned or received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Casting (Active Comparator): Subjects will be treated with serial casting
  Interventions: Procedure: Casting
- Bracing (Active Comparator): Subjects will be treated with full-time orthotics (braces)
  Interventions: Device: Bracing

INTERVENTIONS:
Procedure: Casting — Use of casts applied using corrective maneuvers
  Arms: Casting
Device: Bracing — Use of full-time spinal orthosis
  Arms: Bracing

SUMMARY:
Comparison of casting and bracing for the treatment of idiopathic early onset scoliosis

DETAILED DESCRIPTION:
This study uses a multicenter, prospective hybrid research design, which will combine two methods of treatment assignment (randomized and parent preference) and an embedded internal pilot study for sample size re-estimation. Patients will be treated either with serial casts or a full-time brace and followed until curve resolution, failure or palliation (neither resolution nor failure after 2 years of treatment). Results of this study will provide clinicians and families with evidence to support informed treatment decisions.

ELIGIBILITY:
Will enroll both patients with scoliosis and 1 of their parents/guardians

Inclusion Criteria:

Patient Inclusion

* Diagnosis of idiopathic early-onset scoliosis
* Child standing independently but not older than 3 years of age
* 20≤ Cobb angle ≤70° (largest structural curvature)
* Rib-vertebral angle difference (RVAD) greater than 20 degrees or Rib Phase II
* Parental consent to participate

Parent Inclusion

* Parent or guardian of the minor subject
* Consent to participate
* Able to complete surveys

Exclusion Criteria:

Patient Exclusion

* Previous operative or non-operative treatment for idiopathic early-onset scoliosis
* Not independently walking by 18 months of age or other signs/symptoms indicative of developmental delay

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Curve Response | on or before 24 months of treatment
  Resolution - curve improvement to <15 degrees (as measured on 2 consecutive radiographs)
  Failure
  1. Initial Cobb 20-50° (inclusive): curve progression of ≥20° resulting in a curve ≥50°
  2. Initial Cobb >50°: curve progression of ≥20°
  Palliation - 2 years of treatment without resolution or failure

SECONDARY OUTCOMES:
Patient Health-related Quality of Life (HRQOL) | on or before 24 months of treatment
  Evaluation of patients' HRQOL as estimated by serial administrations of the Early Onset Scoliosis Questionnaire (EOSQ-24, completed by the parent at baseline and every 6 months, total score range 0-100, higher scores indicate higher level of HRQOL). Within and between treatment arm comparisons will be made.

OTHER OUTCOMES:
Parent and Family Functioning | on or before 24 months of treatment
  Evaluation of patients' disease and treatment on parent and family function as estimated by serial administrations of the PedsQL Family Impact Module scores (PedsQL FIM, completed by the parent, total score range 0-100, higher scores indicate less negative impact). Within and between treatment arm comparisons will be made.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart L Weinstein, MD, Principal Investigator — University of Iowa
Locations (26):
- United States (24):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours/Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Shriners Hospitals for Children - Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins, Baltimore, Maryland
  - Children's Hospital of Boston, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - Children's Mercy Kansas City, Kansas City, Missouri
  - St. Louis Children's Hospital/Washington University, St Louis, Missouri
  - Golisano Children's Hospital/University of Rochester, Rochester, New York
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Doernbecher Children's Hospital / OHSU, Portland, Oregon
  - Shriners Hospitals for Children - Portland, Portland, Oregon
  - Children's Hospital of Pennsylvania, Philadelphia, Pennsylvania
  - Shriners Hospitals for Children - Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Italian Scientific Spine Institute (ISICO), Milan, Italy
- Starship Child Health, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
All study data (assessments and images) will reside in the Pediatric Spine Registry.
Supporting Information: Study Protocol
Time Frame: after our planned analyses and publications are completed
Access Criteria: Study data will be available to all CVBT investigators and Pediatric Spine Registry participants. Interested parties will prepare a proposal for consideration by the PI and the Pediatric Spine Study Group. If approved, the Pediatric Spine Registry staff will query the database and provide the required data for secondary analysis.